CLINICAL TRIAL: NCT07165678
Title: A Multi-Centre, Randomised Trial Assessing the Value of Computed Tomography Coronary Angiography Prior to Invasive Coronary Angiography in Patients With Previous Coronary Artery Bypass Grafts in Reducing Cardiac Events
Brief Title: CTCA Prior to Invasive Angiography in Post-Bypass Patients (BYPASS CTCA 2)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 341412; NIHR207209 (Other Grant/Funding Number: NIHR Research for Patient Benefit); PR2300245 (Other Grant/Funding Number: Siemens Healthcare Limited)
Record Dates: First submitted 2025-08-15; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Artery Bypass Graft; Angina; Coronary Artery Disease; CABG; percutaneous coronary intervention; coronary angiograms; Computerised Tomography Coronary Angiography; CTCA
MeSH Terms: conditions — Coronary Disease; Angina Pectoris; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Arm A: coronary angiography alone Arm B: CTCA scan with or without angiography
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICA only (No Intervention): Invasive coronary angiogram (ICA) performed only.
- CTCA with or without ICA (Active Comparator): Computed Tomography Cardiac Angiography (CTCA) with or without invasive coronary angiogram (ICA)
  Interventions: Diagnostic Test: CTCA

INTERVENTIONS:
Diagnostic Test: CTCA — Computed Tomography Cardiac angiography (CTCA) performed prior to invasive coronary angiogram (ICA).
  Other Names: Computed Tomography Cardiac angiography
  Arms: CTCA with or without ICA

SUMMARY:
The goal of this clinical trial is to evaluate whether a coronary computed tomography angiography (CTCA)-guided strategy can reduce the risk of death, heart attack, stroke, and hospital admissions in patients experiencing angina or myocardial infarction following coronary artery bypass graft (CABG) surgery. The main questions it aims to answer are:

* Can CTCA reduce major adverse cardiovascular events compared to standard invasive coronary angiography?
* Is CTCA a cost-effective and safer alternative that improves patient quality of life? Researchers will compare outcomes between patients receiving CTCA prior to angiography and those undergoing standard angiography alone to determine if CTCA improves clinical outcomes and procedural safety.

Participants will:

* Be randomly assigned to either CTCA-guided care or standard angiography
* Undergo coronary imaging and follow-up assessments
* Complete questionnaires on quality of life and healthcare resource use

DETAILED DESCRIPTION:
Patients with prior coronary artery bypass graft (CABG) surgery frequently present with recurrent angina or acute coronary syndromes due to progressive native coronary artery disease or graft failure. Invasive coronary angiography remains the standard diagnostic approach but is technically challenging in this population due to variable graft anatomy, leading to prolonged procedure times, increased radiation exposure, higher contrast volumes, and elevated risk of procedural complications.

Computed Tomography Coronary Angiography (CTCA) offers a non-invasive alternative with high diagnostic accuracy for graft patency and coronary anatomy. Prior observational data (e.g., BYPASS-CTCA study) suggest that CTCA performed prior to invasive angiography may improve procedural efficiency and safety. However, whether CTCA can guide clinical decision-making to avoid unnecessary angiography and improve long-term outcomes remains unproven.

This multi centre, randomised controlled trial will enrol 1,000 patients with prior CABG presenting with angina or myocardial infarction. Participants will be randomised to either a CTCA-guided strategy or standard care involving direct invasive coronary angiography. In the CTCA arm, angiography may be deferred if CTCA findings support medical management. The primary outcome is the composite rate of major adverse cardiovascular events (MACE), including death, myocardial infarction, stroke, and hospitalisation for unstable angina. Secondary outcomes include procedural metrics, patient-reported quality of life, cost-effectiveness, and healthcare resource utilization.

Clinical data will be collected through patient questionnaires, procedural records, and central registry downloads. The study incorporates patient and public involvement throughout its design and implementation. Results will be disseminated via peer-reviewed publications, public-facing reports, and digital platforms.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18
* Previous coronary artery bypass grafting (CABG)
* An indication for coronary angiography

  * Angina
  * Ischaemia on perfusion imaging
  * Acute coronary syndrome
* Patients are able and willing to give their written informed consent

Exclusion Criteria:

* Subjects presenting with ST segment myocardial infarction within window for primary PCI
* Patients considered unsuitable to participate by the research team (e.g. due to medical reasons, laboratory abnormalities, or subject's unwillingness to comply with all study related procedures)
* Life expectancy less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Composite major adverse cardiovascular events (MACE): all-cause mortality, non-fatal stroke, non-fatal myocardial infarction, and cardiovascular hospitalisation | Up to 2.5 years post-randomisation (median follow-up: 18 months)
  Clinical events will be assessed from randomisation until the final patient completes 6 months of follow-up. The composite endpoint includes all-cause mortality, non-fatal stroke, non-fatal myocardial infarction, and cardiovascular hospitalisation. Based on a 2-year recruitment period, individual follow-up will range from 0.5 to 2.5 years, with an estimated median follow-up of 18 months.

SECONDARY OUTCOMES:
Fluoroscopy time during coronary angiography | During coronary angiography procedure
  Unit of Measure: Minutes
Incidence of procedural complications during coronary angiography | During coronary angiography procedure
  Unit of Measure: Number of participants with event
Radiation dose during coronary angiography | During coronary angiography procedure
  Unit of Measure: Milligray (mGy)
Contrast dose administered during coronary angiography | During coronary angiography procedure
  Unit of Measure: Milliliters (mL)
Procedural duration during coronary angiography | During coronary angiography procedure
  Unit of Measure: Minutes Unit of Measure: Milliliters (mL)
Health-related quality of life (EQ-5D-5L) | Baseline, 6 months, 12 months, 18 months, and 24 months
  Assessed using the EQ-5D-5L questionnaire at baseline and every 6 months during follow-up.
Cost-effectiveness and productivity loss | Baseline and every 6 months during follow-up
  Evaluated using patient questionnaires capturing healthcare resource use and productivity loss at baseline and every 6 months.
Days alive and out of hospital | From randomisation until end of follow-up (up to 2.5 years)
  Total number of days the participant is alive and not admitted to hospital during the follow-up period.
  Unit of Measure: Days
Length of hospital stay | From randomisation until end of follow-up (up to 2.5 years)
  Cumulative duration of hospital admissions during the follow-up period Unit of Measure: Days
Major Adverse Cardiovascular Events (MACE) - Individual components | From randomisation until end of follow-up (up to 2.5 years)
  Cumulative duration of hospital admissions during the follow-up period Unit of Measure: Number of events
Composite two-point MACE (death and MI) | From randomisation until end of follow-up (up to 2.5 years)
  Includes death and myocardial infarction as a simplified composite cardiovascular endpoint.
Major Adverse Cardiovascular Events (MACE) - Cumulative incidence | From randomisation until end of follow-up (up to 2.5 years)
  Total number of MACE events per participant during the follow-up period. Unit of Measure: Number of events
Unplanned revascularisation | From randomisation until end of follow-up (up to 2.5 years)
  Number of unplanned coronary revascularisation procedures performed during follow-up.
  Unit of Measure: Number of procedures
Cardiovascular imaging utilisation | From randomisation until end of follow-up (up to 2.5 years)
  Number and type of cardiovascular imaging procedures performed during follow-up.
  Unit of Measure: Number of procedures

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jones, MRCP, PhD, Principal Investigator — Queen Mary University of London

IPD SHARING:
Plan to Share IPD: Yes
Data sharing available from corresponding author upon reasonable request and with approval from trial steering committee.
Supporting Information: Study Protocol
Time Frame: 2028
Access Criteria: Freely available via journal